CLINICAL TRIAL: NCT07215338
Title: Understanding and Mitigating Delayed Onset Muscle Soreness (DOMS)
Brief Title: Effects of Palmar Cooling on the Human Immune System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Wu Tsai Human Performance Alliance (Unknown)
Responsible Party: Principal Investigator, H Craig Heller, Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 73909
Record Dates: First submitted 2025-10-08; First posted 2025-10-10 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Human Immune Response
Keywords: Palmar Cooling; Human Immunology; Exercise Immunology

STUDY DESIGN:
Intervention Model Description: Control arm has palmar temperature device set to 30 degrees celsius, interventional arm has palmar temperature device set to 14 degrees celsius.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 30 degree celsius (Placebo Comparator): Participants will be asked to complete 10 sets of bicep curls to muscle failure with 3 minute rests between sets. The placebo participants will put their palms on a water perfused pad between sets and following the last set. The pads will be perfused with 30 degree C water.
  Interventions: Other: Muscle Temperature Control
- 14 degree celsius (Experimental): Participants will be asked to complete 10 sets of bicep curls to muscle failure with 3 minute rests between sets. For the experimental participants they will rest their palms on a water perfused pad during each 3 minute rests and also following the last set of curls. The pads will be perfused with 12 - 14 degrees Centigrade water. curls to muscle failure.Participants will use the palmar temperature control device set to 14 degree celsius for 3 minutes. between 10 sets of bicep curls matched to control counterpart.
  Interventions: Other: Muscle Temperature Control

INTERVENTIONS:
Other: Muscle Temperature Control — The intervention will be placing the palms of the hands on a water perfused pad.

SUMMARY:
This is a research study on human exercise that will investigate the immune system response post-exercise and how it relates to Delayed Onset Muscle Soreness (DOMS), and possible causes for DOMS.

Blood draws (10mL) will be obtained at 5 timepoints: Baseline before intervention, day of exercise immediately following exercise, and post-exercise days 1, 2 and 4.

Point of care lactate levels obtained before and after exercise.

Subjective pain scores recorded daily starting immediately after after exercise.

ELIGIBILITY:
Inclusion Criteria:

- Ability to perform two arm bicep curl of at least 35 lb as 1 repetition maximum

Exclusion Criteria:

* Autoimmune disease
* Steroid use
* On current immune-modifying treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2024-06-28 (Actual); Primary Completion 2024-09-27 (Actual); Study Completion 2024-09-27 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in phosphorylation markers in the Janus kinase/signal transducer and activator of transcription (JAK/STAT) and Toll-like Receptor (TLR)-pathway in immune cell populations | From enrollment to 5 days after the end of treatment
  Collected at baseline from whole blood prior to exercise, day of exercise, post-exercise day 1, post-exercise day 2, post-exercise day 4

SECONDARY OUTCOMES:
Change from pre-exercise baseline in point of care lactate levels | 1 day
  Two point of care lactate draws before and after exercise obtained in mmol/L
Change in Pain Scores from baseline | From day of intervention daily for 5 days.
  Daily subjective pain scores recorded according to the Borg Perceived Pain Scale from 0 (no pain) to 11 (maximum pain)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Tsai, MD, Study Director — Stanford University; Brice Gaudilliere, MD, PhD, Principal Investigator — Stanford University; H. Craig Heller, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Age, Sex, Biological information
Supporting Information: Study Protocol
Time Frame: Data is available now and will remain available.
Access Criteria: Access through RedCap

REFERENCES:
- [Background] Grahn DA, Cao VH, Heller HC. Heat extraction through the palm of one hand improves aerobic exercise endurance in a hot environment. J Appl Physiol (1985). 2005 Sep;99(3):972-8. doi: 10.1152/japplphysiol.00093.2005. Epub 2005 May 5. PMID 15879169